CLINICAL TRIAL: NCT04765202
Title: A Phase 1/2a, Controlled, Randomized, Multicenter Study Evaluating the Efficacy, Safety, and Tolerability of StrataGraft Overlay of Meshed Autograft (SOMA) in Treatment of Full-Thickness Thermal Burns
Brief Title: StrataGraft Overlay of Meshed Autograft in Full-thickness Thermal Burns
Acronym: StrataSOMA
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business Reason
Sponsor: Stratatech, a Mallinckrodt Company (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MNK01062117
Record Dates: First submitted 2021-02-04; First posted 2021-02-21 (Actual); Results first posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Full Thickness Thermal Burn

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort1 Group1: AG Tx Sites (Experimental): Participants received autograft treatment (AG Tx) consisting of autograft alone (mesh ratio "m", per clinical judgment) at the treatment site on Day 1.
  Interventions: Procedure: AG Tx
- Cohort1 Group1: SOMA Tx Sites (Experimental): Participants received StrataGraft overlay of meshed autograft (SOMA Tx) at the treatment site in which m+1:1 meshed autograft was overlaid with StrataGraft, and applied to wounds of 100 to 400 square centimeters (cm^2) in area on Day 1.
  Interventions: Biological: SOMA Tx
- Cohort1 Group 2: AG Tx Sites (Experimental): Participants received AG Tx consisting of autograft alone (mesh ratio "m", per clinical judgment) at the treatment site on Day 1.
  Interventions: Procedure: AG Tx
- Cohort1 Group2: SOMA Tx Sites (Experimental): Participants received SOMA Tx on the treatment site in which m+2:1 meshed autograft was overlaid with StrataGraft, and applied to wounds of 100 to 400 cm^2 in area on Day 1.
  Interventions: Biological: SOMA Tx

INTERVENTIONS:
Procedure: AG Tx — Control treatment that is meshed autograft alone applied to a burn area.
  Other Names: Meshed Autograft
  Arms: Cohort1 Group 2: AG Tx Sites; Cohort1 Group1: AG Tx Sites
Biological: SOMA Tx — Meshed autograft applied to the burn area and covered with StrataGraft.
  Other Names: StrataGraft skin tissue Overlay of Meshed Autograft (SOMA)
  Arms: Cohort1 Group1: SOMA Tx Sites; Cohort1 Group2: SOMA Tx Sites

SUMMARY:
Autografting is a surgical procedure to transplant healthy skin (donor skin) from another part of the participant's own body (donor site) to the burned part. Autografting is the usual treatment for full-thickness (FT) burns.

It works to close the wound, but can cause other problems:

* Donor sites are painful, can become infected or scarred, or can even become FT wounds themselves
* Treatment problems can require more grafting
* Additional surgery increases risk of medical problems caused by the treatment

Stratatech is trying to find a safe and effective treatment option for severe burns that uses less donor skin.

All participants in this study received meshed autograft on one part of their burn (AG Tx). They received more widely meshed than AG Tx site autograft with a StrataGraft covering (SOMA Tx) on a different part of their burn.

ELIGIBILITY:
Inclusion Criteria:

* Has 2% to 49% (inclusive) total body surface area (TBSA) thermal burn area, including areas of full thickness (FT) injury clinically indicated for surgical excision and autografting, appropriate for protocol-defined treatment areas
* Meets protocol-specified criteria for qualification and contraception
* Is willing and able to comply with all study procedures and requirements
* Voluntarily consents to participate and provides written informed consent prior to any protocol-specific procedures

Exclusion Criteria:

* Is a prisoner, pregnant, or had previous autografting to treatment sites
* Is expected to survive less than 3 months
* Is participating in another interventional trial, or did within 30 days before enrollment
* Has anticipated treatment sites that are outside protocol-specified parameters
* Has concurrent clinically significant inhalation injury, inadequate fluid resuscitation, or burns of chemical or electrical (non-thermal) etiology
* Has other signs, symptoms or history of any condition that, per protocol or in the opinion of the investigator, might compromise:

  1. The safety or well-being of the participant
  2. The study objectives

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team Leader, Study Director — Stratatech, a Mallinckrodt Company
Locations (5):
- United States (5):
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Tampa General Hospital / University of South Florida, Tampa, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Stony Brook University, Stony Brook, New York
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 5 investigative sites in the United States from 10 October 2021 to 07 June 2024.
Pre-assignment Details: The study was planned to be conducted in 2 cohorts. Only Cohort 1 data is reported, as the study was terminated before any participant was enrolled in Cohort 2. Total 13 participants were randomized in Cohort 1, each participant served as their own control. All participants had 2 treatment sites that were randomized to receive autograft treatment (AG Tx) at 1 treatment site, and StrataGraft overlay of meshed autograft (SOMA Tx) on the 2nd treatment site.
Units Other Than Participants: treatment sites
Groups:
- Cohort1 Group1: AG Tx: Participants who received AG Tx consisting of autograft alone (mesh ratio "m", per clinical judgment) at the treatment site on Day 1.
- Cohort1 Group1: SOMA Tx: Participants who received SOMA Tx at the treatment site in which m+1:1 meshed autograft was overlaid with StrataGraft, and applied to wounds of 100 to 400 square centimeters (cm^2) in area on Day 1.
- Cohort1 Group2: AG Tx: Participants received AG Tx consisting of autograft alone (mesh ratio "m", per clinical judgment) at the treatment site on Day 1.
- Cohort1 Group2: SOMA Tx: Participants received SOMA Tx on the treatment site in which m+2:1 meshed autograft was overlaid with StrataGraft, and applied to wounds of 100 to 400 cm^2 in area on Day 1.
Period: Overall Study
Arm/Group | Cohort1 Group1: AG Tx | Cohort1 Group1: SOMA Tx | Cohort1 Group2: AG Tx | Cohort1 Group2: SOMA Tx
Started | 7; 7 treatment sites | 7; 7 treatment sites | 6; 6 treatment sites | 6; 6 treatment sites
Completed | 6; 6 treatment sites | 6; 6 treatment sites | 3; 3 treatment sites | 3; 3 treatment sites
Not Completed | 1; 1 treatment sites | 1; 1 treatment sites | 3; 3 treatment sites | 3; 3 treatment sites
Not completed — Lost to Follow-up | 1 | 1 | 2 | 2
Not completed — Physician Decision | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all participants who were randomized and treated with at least one area of SOMA Tx and one area of AG Tx.
Groups:
- Cohort 1 Group 1: Participants received AG Tx consisting of autograft alone (mesh ratio "m", per clinical judgment) at 1 treatment site compared to SOMA Tx on other treatment site in which m+1:1 meshed autograft was overlaid with StrataGraft, applied to wounds of 100 to 400 cm^2 in area on Day 1.
- Cohort 1 Group 2: Participants received AG Tx consisting of autograft alone (mesh ratio "m", per clinical judgment) at treatment site compared to SOMA Tx on other treatment site in which m+2:1 meshed autograft was overlaid with StrataGraft, applied to wounds of 100 to 400 cm^2 in area on Day 1.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Group 1 | Cohort 1 Group 2 | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (12.20) | 47.2 (12.54) | 47.3 (11.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 7 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 4 | 8
  Black or African American | 1 | 0 | 1
  Not Reported | 1 | 2 | 3
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Sites With Complete Wound Closure Without Additional Autografting at Month 2
Description: Confirmed complete wound closure was defined as complete skin re-epithelialization without drainage confirmed at 2 visits at least 2 weeks apart but no later than Week 20. Complete wound closure was considered to have occurred at the earlier of the 2 observations of complete skin re-epithelialization without drainage. The number of treatment sites with complete wound closure without additional autografting at Month 2 was reported.
Time Frame: At Month 2
Population: FAS included all participants who were randomized and treated with at least one area of SOMA Tx and one area of AG Tx.
Measure: Number; unit: treatment sites
Units Other Than Participants: sites
Groups:
- Cohort1 Group1: SOMA Tx: Participants who received SOMA Tx at the treatment site in which m+1:1 meshed autograft was overlaid with StrataGraft, and applied to wounds of 100 to 400 cm^2 in area on Day 1.
Arm/Group | Cohort1 Group1: AG Tx | Cohort1 Group1: SOMA Tx | Cohort1 Group2: AG Tx | Cohort1 Group2: SOMA Tx
Number analyzed (Participants) | 7 | 7 | 6 | 6
Number analyzed (sites) | 7 | 7 | 6 | 6
treatment sites | 6 | 7 | 6 | 6
Statistical Analysis 1: Comparison: Cohort1 Group1: AG Tx vs Cohort1 Group1: SOMA Tx; Comparison of complete wound closure without additional autografting at Month 2 in AG TX site and SOMA TX site in Cohort 1 Group 1; Test type: Superiority; p = 1.0000, Fisher Exact; Percentage Difference = 14.3, 95% CI 2-sided [-11.64 to 40.21] — Difference was calculated as (percent area of wound closure in SOMA Tx site) - ((percent area of wound closure in AG Tx site). 95% CI was derived using the normal approximation to binomial distribution
Statistical Analysis 2: Comparison: Cohort1 Group2: AG Tx vs Cohort1 Group2: SOMA Tx; Comparison of complete wound closure without additional autografting at Month 2 in AG TX site and SOMA TX site in Cohort 1 Group 2; Test type: Superiority; Percentage Difference = 0, 95% CI 2-sided [0 to 0] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Number of Participants With Durable Wound Closure of Study Treatment Sites Without Additional Autografting at Month 12
Description: Durable wound closure is defined as persistence of closure, maintained for at least 3 months after the initial observation of closure.
Time Frame: At Month 12
Population: FAS included all participants who were randomized and treated with at least one area of SOMA Tx and one area of AG Tx. Here, the overall number analyzed of participants are the number of participants with data available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Group 1 | Cohort 1 Group 2
Number analyzed (Participants) | 6 | 3
Participants
  AG Tx Site | 6 | 3
  SOMA Tx Site | 6 | 3

ADVERSE EVENTS:
Time Frame: Up to 13 months
Description: Safety population included all participants who signed the informed consent form (ICF) and were treated with the investigational treatment.
Groups:
- Cohort 1 Group 1: All Participants: Participants received AG Tx consisting of autograft alone (mesh ratio "m", per clinical judgment) at 1 treatment site compared to SOMA Tx on other treatment site in which m+1:1 meshed autograft was overlaid with StrataGraft, applied to wounds of 100 to 400 cm^2 in area on Day 1.
- Cohort 1 Group 1: AG Tx Sites: Participants who received AG Tx consisting of autograft alone (mesh ratio "m", per clinical judgment) at the treatment site on Day 1.
- Cohort 1 Group 1: SOMA Tx Sites: Participants who received SOMA Tx at the treatment site in which m+1:1 meshed autograft was overlaid with StrataGraft, and applied to wounds of 100 to 400 cm^2 in area on Day 1.
- Cohort 1 Group 2: All Participants: Participants received AG Tx consisting of autograft alone (mesh ratio "m", per clinical judgment) at treatment site compared to SOMA Tx on other treatment site in which m+2:1 meshed autograft was overlaid with StrataGraft, applied to wounds of 100 to 400 cm^2 in area on Day 1.
- Cohort 1 Group 2: AG Tx Sites: Participants received AG Tx consisting of autograft alone (mesh ratio "m", per clinical judgment) at the treatment site on Day 1.
- Cohort 1 Group 2: SOMA Tx Sites: Participants received SOMA Tx on the treatment site in which m+2:1 meshed autograft was overlaid with StrataGraft, and applied to wounds of 100 to 400 cm^2 in area on Day 1.
Arm/Group | Cohort 1 Group 1: All Participants | Cohort 1 Group 1: AG Tx Sites | Cohort 1 Group 1: SOMA Tx Sites | Cohort 1 Group 2: All Participants | Cohort 1 Group 2: AG Tx Sites | Cohort 1 Group 2: SOMA Tx Sites
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/7 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/7 | 0/7 | 1/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 7/7 | 3/7 | 1/7 | 6/6 | 3/6 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Group 1: All Participants (N=7) | Cohort 1 Group 1: AG Tx Sites (N=7) | Cohort 1 Group 1: SOMA Tx Sites (N=7) | Cohort 1 Group 2: All Participants (N=6) | Cohort 1 Group 2: AG Tx Sites (N=6) | Cohort 1 Group 2: SOMA Tx Sites (N=6)
Homicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Group 1: All Participants (N=7) | Cohort 1 Group 1: AG Tx Sites (N=7) | Cohort 1 Group 1: SOMA Tx Sites (N=7) | Cohort 1 Group 2: All Participants (N=6) | Cohort 1 Group 2: AG Tx Sites (N=6) | Cohort 1 Group 2: SOMA Tx Sites (N=6)
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pilonidal cyst (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Vascular device infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Exposure to communicable disease (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Skin graft failure (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypertrophic scar (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 2 | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Blood pressure diastolic abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-09-28): https://cdn.clinicaltrials.gov/large-docs/02/NCT04765202/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-26): https://cdn.clinicaltrials.gov/large-docs/02/NCT04765202/SAP_001.pdf